CLINICAL TRIAL: NCT04258215
Title: PSA Extraglottic Airway for Positive Pressure Ventilation (Pharachute Supralaryngeal Airway)
Brief Title: PSA (Pharachute Supralaryngeal Airway) for Positive Pressure Ventilation (PPV)
Acronym: PSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSA device PPV study
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Airway Control
Keywords: Positive pressure ventilation; Extraglottic Airway Device

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive pressure achieved with PSA (Experimental): Maximum airway inflation pressure achievable before a significant leak occurs.
  Interventions: Device: Experimental: Routine positive pressure airway management.

INTERVENTIONS:
Device: Experimental: Routine positive pressure airway management. — The use of the PSA extraglottic airway for routine general anesthesia will be assessed for quality of airway management by measuring the seal pressure when using the device in 20 participants.

SUMMARY:
The Pharachute Supralaryngeal Airway (PSA) is an extraglottic airway device (EAD) for routine use in anaesthesia.

The plan is to do a pilot study on a minimum of 20 and maximum of 30 participants whose fitness status is ASA 1 or 2 for whom this type of airway management is routinely used. When the participants are asleep the airway will be inserted, with ease of insertion and satisfactory positive pressure ventilation assessed. This will be indicated by minimal threshold leak from the breathing system and the seal pressure that can be achieved. Any side-effects will be assessed post-operatively.

DETAILED DESCRIPTION:
The proposed research is non-commercial. No extraglottic airways are good enough to displace the use of tracheal tubes, currently used in 40+% of general anaesthesia. Anaesthesia requiring tracheal tube intubation is associated with 0.1% with permanent voice changes1. That means, 800 people per annum in the UK will suffer permanent voice changes. Reduction of the use of tracheal tubes to 10% will reduce this problem by 600 per annum. The PSA device is a new extraglottic airway designed with the purpose of achieving better sealing pressures safely because of a different sealing site and self-energizing sealing mechanism and a better prevention of the risk of aspiration in the presence of regurgitation. Therefore, it has the potential to make a huge difference to patients. As a first step in this objective, the investigators need to find out whether the airway device is predictably reliable and whether the seal pressures are good enough for positive pressure ventilation.

3. Research hypothesis

The PSA is a reliable extraglottic airway that can be inserted easily, atraumatically and achieves reliable sealing pressures that will allow for positive pressure ventilation.

4. Research questions

Concerning the use of the PSA in general anaesthesia

* How easy is it to insert?
* Is there a placement learning curve?
* What is its maximum sealing pressure?
* What is the usual ventilation pressure
* Severity and incidence of minor postoperative complications such as sore throat, dysphagia, hoarseness etc?

  5. Objectives

5.1 Primary endpoints Ease of insertion - number of attempts

time taken mechanical trauma - is there blood on the device at removal?

Maximum peak inspiratory pressure during manual controlled ventilation. Sealing pressure during controlled ventilation.

5.2 Secondary endpoints

Postoperative complications:

- nausea and vomiting

hoarseness sore throat difficulty swallowing neck pain hearing problems mouth pain

tongue numbness

6. Study design

Participants will be informed as to the side-effect risks about the airway device they are to receive in a manner that compares it with the alternative airway management strategy, which they will be free to choose instead.

The peak airway and sealing pressures will be measured intra-operatively using the pressure gauge on the anaesthetic machine.

The participant will be assessed for postoperative complications. This will take the form of a postoperative questionnaire, which can be found in appendix iii. They will be asked about the complications at 2hrs postoperatively and 24hrs postoperatively.

6.1 Subject selection

The subjects will all be adult ASA (American Society of Anesthesiologists) grade 1-2 participants, who are competent to consent and who are undergoing elective surgical procedures. The ASA grading can be found in the appendix (ii).

6.2 Inclusion criteria

Males and females between 165 and 175 cm height. (This height restriction is because this initial study will be limited to the availability of one size [4] only for this pilot study). The selection of participants for the study may also include the matching of the width of the thyroid cartilage to the width of the PSA.

Age 16-89 inclusive. ASA grade 1-2. Undergoing elective surgery. Able to give written and signed informed consent.

The inclusion criteria may have to change as there is only one size of PSA to test and the investigators are yet to work out whether the above best estimate of how to select the correct size is accurate. So, it would appear to be a logical plan to include in the study design a test to verify the above selection criterion using a maximum of the first 10 participants that may not be included in the study that will be published, unless the above selection criteria is validated, i.e. does not require any adjustment.

6.3 Exclusion criteria

Requiring emergency surgery.

6.4 Sample size

20 participants: Reasons for the choice of this number is based upon other appropriate respective studies both pilot and randomized controlled studies (only 22 and 60 cases in the case of the SLIPA airway2,3) conducted by this author and many other similar studies published in the literature (See literature review). As this is a pilot study, it would seem that the right number the investigators should choose is the minimum number of participants to enable us to answer the primary question reliably, although it is probably too few to give meaningful answer to the the secondary questions. Nevertheless, this data may still be useful and sufficient to exclude unanticipated serious side-effects.

6.5 Informed consent

Participants will be visited as part of the normal preoperative visit, (this will be mainly day surgery, so before the operating list begins). Those who satisfy the inclusion criteria will be approached for the study, given a participant information leaflet to read and time to ask any questions they may have. Informed consent will be obtained prior to the participant undergoing any procedure. . Only a study doctor who has been trained, is competent and is on the study delegation log will participate in the consent process.

The investigator will ask the participant immediately before anaesthesia is induced if they have any further questions and to confirm that they still wish to take part in the study.

7. Study procedure

7. Immediately before day surgery begin

- Discussion of trial.

Provision of information leaflet. Discussion of questions arising from the leaflet.

7.2 In the induction room before anaesthesia commences

Any further questions about the study. The opportunity to change their minds

Verbal confirmation of the signed informed consent.

8. Anaesthetic induction and maintenance No special test equipment is needed for this study other than what is in everyday current use.

Standard monitoring to be attached before induction. Anaesthesia induction with 1mcg/kg fentanyl and 1-3mg/kg propofol to loss of verbal contact.

Neuromuscular relaxation, only if required by the surgery, including the use of twitches on Train of Four monitoring (TOF).

Anaesthesia maintained with Sevoflurane in an air/oxygen mixture.

9. Insertion of PSA device According to manufacturer's insertion guidelines (participant must be deep enough or muscle relaxant working according to TOF).

Time for insertion from picking up device to attachment of breathing system measured.

Number of attempts documented.

* 10. Adequacy of ventilation Manual ventilation immediately following insertion. Adequacy of chest wall movement, end tidal carbon dioxide waveform noted. If repositioning required then intervention (head extension, neck flexion, jaw thrust) and effect noted.

If ventilation is unsatisfactory following two insertions of the medical device this will be abandoned and alternative airway management instituted.

11. Positive pressure ventilation Target tidal volume of 6mL/kg (milliliters per kilogram). Ratio of Inspiration: Expiration between 1:1 and 1:2.

Set rate adjusted to maintain end tidal carbon dioxide 4 - 5 kiloPascals (kPa).

12. Measurement of airway pressures

12.1 Peak airway pressure

- At steady state

12.2 Seal pressure

Spill valve occlusion. Seal pressure regarded as that pressure at which gas heard to be leaking from around the sealing flange of the device (Manual pressure control by squeezing the bag may be used to achieve this rapidly, thus minimizing the time period of application of the Valsalva manoeuvre effect [peak pressure less than two seconds], thus minimizing risk to the participant as regards effect upon the cardiovascular system (CVS) and barotrauma).

Limited to a maximum of 40cm water pressure.

13. Removal of device Once surgery completed. Anaesthesia discontinued, TOF 1:4 > 75% and reversal agent if appropriate.

Removal of device once participant able to open eyes and mouth to command.

14. Postoperative follow up

Participants will be asked to complete a postoperative questionnaire (Appendix iii) at the following time points:

2hrs postoperatively (when the participant will still be in the Recovery Ward)

24hrs postoperatively Any complications that last up to 24 hours and are more than just mild and fading symptoms will be considered serious enough to necessitate the patient being seen again as soon as possible and assessed as to the need for treatment or referral to a general practitioner for management. This will also immediately trigger consideration as to whether to discontinue the trial and the product development.

References:

Yamanaka H et al Brit. J. Anaesthesia 103(3):452-5 (2009) 3093 participants prospectively studied. Arytenoid dislocation 1:1000.

2 Miller D M, Lavelle M. A Streamlined Pharynx Airway Liner: Pilot Study in 22 Participants in Controlled and Spontaneous Ventilation, Anesthesia Analgesia 2002;94:759-761.

3. Miller D M, Light D. Laboratory and clinical comparisons of the Streamlined Liner of the Pharynx Airway (SLIPA™) with the laryngeal mask airway. Anaesthesia 2003; 58: 136-142.

ELIGIBILITY:
Inclusion Criteria:

* Anatomical sizing criterion

Exclusion Criteria:

* Emergency participants Suspected full stomach
* Mentally incompetent patients
* Patients who are requiring head and neck surgery
* Morbidly obese patients

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
1.PSA Ease of insertion It should be adequate and reliable [Time Frame: Assessed by the anesthesiologist within first 60 seconds of inserting the device.] | Assessed by the anesthesiologist within first 60 seconds of inserting the device.
  Time taken to achieve adequate airway
Satisfactory positive pressure ventilation: Maximum airway inflation pressure | Assessed by the anesthesiologist within first 120 seconds of inserting the device.
  Maximum airway inflation pressure that can be achieved before a significant leak becomes apparent must exceed 14 cm water pressure.

SECONDARY OUTCOMES:
Watching for possible unanticipated serious side effects from airway usage | Within the first 24 hours
  Sore throat, bleeding, voice changes, swallowing difficulty, localized neurological damage.

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Pai, Principal Investigator — Hull University Teaching Hospital NHS Trust; Donald Miller, Study Director — Hull University Teaching Hospital NHS Trust
Locations (1):
- Hull University Teaching Hospital, Castle Hill Hospital., Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller DM, Light D. Laboratory and clinical comparisons of the Streamlined Liner of the Pharynx Airway (SLIPA) with the laryngeal mask airway. Anaesthesia. 2003 Feb;58(2):136-42. doi: 10.1046/j.1365-2044.2003.02962.x. PMID 12562409
- [Result] Yamanaka H, Hayashi Y, Watanabe Y, Uematu H, Mashimo T. Prolonged hoarseness and arytenoid cartilage dislocation after tracheal intubation. Br J Anaesth. 2009 Sep;103(3):452-5. doi: 10.1093/bja/aep169. Epub 2009 Jun 25. PMID 19556269
- [Result] Miller DM, Lavelle M. A streamlined pharynx airway liner: a pilot study in 22 patients in controlled and spontaneous ventilation. Anesth Analg. 2002 Mar;94(3):759-61; table of contents. doi: 10.1097/00000539-200203000-00052. PMID 11867412